CLINICAL TRIAL: NCT03766672
Title: Characterization of the Genetic Profile of Type 2 Endometrial Carcinoma in Martinique
Acronym: ENDO-NGS-MQ
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Martinique Cancer Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH2_15; 2018-A02091-54 (Other: ANSM)
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Neoplasms
Keywords: Endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples for extraction of DNA on whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention Arm: Identify the genetic profile of type 2 endometrial carcinomas in Martinique from tumor sample for extraction of tumor DNA .
  Interventions: Diagnostic Test: Intervention Arm

INTERVENTIONS:
Diagnostic Test: Intervention Arm — The intervention consists to the characterization of molecular mechanisms using to Next Generation Sequencing (NGS) technique.

SUMMARY:
In Martinique, about 33 new cases are diagnosed per year, with a high incidence rate of type 2 endometrial carcinoma which has a poor prognosis with few therapeutic options. Although targeted therapies are used in many types of cancer, they are still possible a minority of patients. In current practice, endometrial cancers do not benefit these therapies. Characterization of the molecular mechanisms involved in the genesis of type 2 endometrial carcinoma could help to identify biomarkers predictive of a response to targeted therapies. We propose to identify the genetic profile of type 2 endometrial carcinomas in Martinique.

DETAILED DESCRIPTION:
Type 2 endometrial carcinomas are often diagnosed at advanced stages, with an high risk of metastatic recurrence and death even when diagnosed at early stages. They also have few therapeutic options. The Characterize the mutations responsible of cancer development has led to develope "precision medicine" that targets "actionable genes" by a drug. This concept of actionable mutation refers to a change in the DNA molecule that can predict the response to a drug defined as targeted therapy. Although targeted therapies are used in many types of cancer, they still target a minority of patients. Some tumor sites still do not benefit from these treatments. Specifically, type 2 endometrial cancers that have poor prognosis with few therapeutic options. The characterization of molecular mechanisms, by Next Generation Sequencing (NGS), involved in the carcinogenesis of endometrial cancers, particularly type 2 cancers, should allow the identification of predictive biomarkers for response to certain targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Major subject living in Martinique with the following characteristics :

  * Patients with type 2 endometrial cancer, with anatomopathological confirmation
  * Affiliate or beneficiary of french social security.
  * Free, informed with a written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any research required by the research).

Exclusion Criteria:

* Type 1 adenocarcinoma
* Patients not affiliated to french social security
* Refusal to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women aged more 18 years living in Martinique with a type 2 endometrial cancer confrimed by with anatomopathological reports.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Number of biomarkers identified by Next Generation Sequencing involved in type 2 endometrial tumors in Martinique | 24 Months
  Characterization of potentially operable mutations in type 2 endometrial tumors from DNA sample withdraw at inclusion and during follow visit

CONTACTS AND LOCATIONS:
Overall Officials: Medhi JEAN-LAURENT, MD, Principal Investigator — CHU Martinique
Locations (1):
- Chu Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No